CLINICAL TRIAL: NCT05596890
Title: Patient-reported Outcome-based Surveillance System Evaluating Safety and Efficacy of Preoperative Immunochemotherapy +/- Chemoradiation in Patients With Esophageal Squamous Cell Carcinoma - A Prospective, Explorative, Phase II Study
Brief Title: Patient-reported Outcomes in Preoperative Immunochemotherapy/Radiotherapy-treated Esophageal Cancer Patients
Acronym: PICCRT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RICE-PICCRT
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Esophageal Squamous Cell Carcinoma; Patient-reported Outcomes; Immunotherapy
Keywords: Pathological complete response; Efficacy; Safety; Dysphagia
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Deglutition Disorders | interventions — Cisplatin; Carboplatin; tislelizumab; Radiotherapy, Intensity-Modulated; Esophagectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant immunochemotherapy +/- short-term radiotherapy (Experimental): Tislelizumab + cisplatin/carboplatin + albumin-bounded paclitaxel +/- radiotherapy
  Interventions: Drug: Paclitaxel-albumin; Drug: Cisplatin; Drug: Carboplatin; Drug: Tislelizumab; Radiation: VMAT or IMRT; Procedure: Esophagectomy

INTERVENTIONS:
Drug: Paclitaxel-albumin — 260mg/m2, ivdrip, d1
Drug: Cisplatin — 60mg/m2, ivdrip, d1
Drug: Carboplatin — AUC=4-6, ivdrip, d1
Drug: Tislelizumab — 200mg, ivdrip, d1
Radiation: VMAT or IMRT — 15Gy/5F (d43-d50, d57-d64), 5 times a week
Procedure: Esophagectomy — Minimally-invasive or open McKeown and Ivor-Lewis esophagectomy

SUMMARY:
Preoperative Immune checkpoint inhibitors combined with chemotherapy have revolutionized the treatment landscape of locally advanced esophageal squamous cell carcinoma. However, there are still a significant proportion of patients who could not benefit from such treatment modality. Currently, no effective biomarkers were identified to stratify responders and non-responders. Early dynamic and persistent relief of dysphagia may act as a predictive biomarker to reflect the on-treatment anti-tumor activity. In this prospective study, we aimed to explore the feasibility of using patient-reported outcomes (PROs) to predict the pathological complete response of esophageal squamous cell carcinoma patients treated with neoadjuvant immunochemotherapy with or without short-term radiation as well as to assess the efficacy and safety of short-term radiotherapy in PROs-insensitive patients after one cycle of neoadjuvant immunochemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed esophageal squamous cell carcinoma
* Potentially resectable esophageal squamous cell carcinoma at first diagnosis (cT1-4aN1-2M0, cT3-T4aN0M0)
* Treatment-naive
* Expected life span > 6 months
* Aged 18 - 75 years old
* Adequate organ functions
* PS 0-2
* Participants are fully informed about the whole study and are willing to sign the informed consent

Exclusion Criteria:

* Previous history of thoracic surgery or radiation
* Cervical or multi-origin esophageal cancer
* Known or suspected experimental drug allergy
* Pregnant or lactating women
* Esophagomediastianl fistula
* Peripheral neuropathy
* Previous cancer history other than esophageal cancer
* Severe organ function deterioration that can not tolerate neoadjuvant therapy
* Previous autoimmune diseases
* diabetic history > 10 years
* interstitial pulmonary disease, non-infectious pulmonitis
* Active type B hepatitis
* Any other conditions that may affect patients' safety and compliance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-30 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response rate | Three to five working days after surgery
  The rate of pathologic complete response rate after the combined treatment of chemotherapy and immunotherapy following surgery

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 24 weeks
  iRECIST criteria defined complete response and partial response
Safety as measured by number of participants with Grade 3 and 4 adverse events | Up to 12 weeks
  Number of Grade 3 and 4 adverse events as defined by CTCAE v5.0
R0 resection rate R0 resection rate R0 resection rate R0 resection rate R0 resection rate R0 resction rate | Three to five working days after surgery
  The R0 resection rate of esophagectomy
Major pathological response | Three to five working days after surgery
  less than 10% residual viable tumor follow neoadjuvant therapy
Overall survival | From the date of diagnosis to the date of death, assessed up to 100 months
  Overall survival rate
Event-free survival | From the date of treatment initiation to the date of first progression (local recurrence of tumor or distant metastasis) or death from any cause, assessed up to 100 months
  EFS
Dysphagia relief score | score calculated by EORTC OES-18 dysphagia scale criteria at each cycle up to 6 months
  DRS

CONTACTS AND LOCATIONS:
Overall Officials: Guibin Qiao, MD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Huang S, Yu H, Li Z, Tang Y, Luo L, Wu J, Li X, Shi Q, Xie S, Qiao G. Electronic patient-reported outcome-based surveillance system to evaluate safety and efficacy of preoperative immunochemotherapy with or without short-term chemoradiation in patients with esophageal squamous cell carcinoma (ePRO-PICCRT): protocol for a prospective, single-arm, phase II study. J Thorac Dis. 2024 Jul 30;16(7):4719-4726. doi: 10.21037/jtd-24-274. Epub 2024 Jul 8. PMID 39144362